CLINICAL TRIAL: NCT00877188
Title: Effect of Combined Aerobic and Resisted Exercise in Breast Cancer Survivors: Upper Extremity Function, Quality of Life and Fitness Outcomes
Brief Title: Effect of Combined Aerobic and Resisted Exercise in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200808034R; NTUH98-M1178
Record Dates: First submitted 2009-03-22; First posted 2009-04-07 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Exercise; Physical Function
Keywords: breast cancer; exercise; upper extremity function; quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise (Experimental): supervised combined aerobic and resistance training for 12 weeks
  Interventions: Other: exercise
- control (No Intervention): waist list control with usual care

INTERVENTIONS:
Other: exercise — supervised combined aerobic and progressive resistance training for 12 weeks
  Arms: exercise

SUMMARY:
The purpose of this study is to evaluate the effects of a combined aerobic and resistance exercise program in breast cancer survivors.

DETAILED DESCRIPTION:
Cancer and cancer treatment side effects are associated with fatigue, pain, decreased cardiovascular fitness and muscle strength, and overall quality of life. Furthermore, cancer survivors are at increased risk for cancer recurrence and for secondary effect such as cardiovascular disease, diabetes, obesity, osteoporosis, and functional decline. Increase physical activity or exercise is proposed to overcome the negative psychological and physiological effects. Preliminary research evidence shows that exercise in cancer survivors improves quality of life, cardiorespiratory fitness, physical functioning, and decrease of fatigue. However, the best exercise mode and intensity has not been well established. Little is known regarding the long term effect. No study investigated impact of exercise for breast cancer survivors on upper extremity function, and correlation between fitness, upper extremity function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* stage 0 to II breast cancer diagnosed within 5 years
* complete adjuvant therapy > 2 months, except hormone therapy
* > 18 years

Exclusion Criteria:

* disease in progress, recurrent, or metastasis
* medical or musculoskeletal condition which resistance exercise is contraindicated
* medication which may alter exercise response

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
muscle fitness, quality of life, upper extremity function | baseline, 12 weeks post exercise training and follow up 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PHD, Study Chair — Graduate School of Physical Therapy, College of Medicine, Nationall Taiwan University, Taipei, Taiwan
Locations (1):
- Graduate School of Physical Therapy, College of Medicine, NTU, Taipei, Taiwan